CLINICAL TRIAL: NCT00233831
Title: Millimeter Wave Therapy (MWT) Versus Placebo for Analgesia and Wound Healing After Elective Total Knee Arthroplasty - a Randomized Controlled Trial
Brief Title: Millimeter Wave Therapy (MWT) for Analgesia After Total Knee Replacement
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: III UV 11/03
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Pain; Acute Pain
Keywords: Postoperative pain; analgesia; total knee arthroplasty
MeSH Terms: conditions — Pain; Acute Pain; Pain, Postoperative; Agnosia

INTERVENTIONS:
Device: Generator of electromagnetic millimeter waves

SUMMARY:
The aim of the study was to test whether the exposure to electromagnetic millimeter waves - Millimeter Wave Therapy (MWT) is effective for relief of acute postoperative pain in patients after elective unilateral total knee arthroplasty (TKA)

ELIGIBILITY:
Inclusion Criteria:

* patients with an American Society of Anesthesiologists physical status of II or III scheduled for elective TKA
* without previous opioid medication
* patients 35-80 years old able to use PCA pumps and Visual Analogue Scale for pain intensity measurement
* patients who have signed consent form

Exclusion Criteria:

* pregnant or nursing females
* recidivist alcoholics
* extremely obese patients (body mass index > 35)
* inability to operate PCA-pump.
* females with the history of unstable angina pectoris (s. Risks for participants)
* patients who are unable to understand the consent form
* systemic infection
* history of psychiatric disease
* necessity to change postoperative analgesic scheme for particular patient
* severe intercurrent disease during the course of MWT

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-03; Primary Completion 2006-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Total amount of weak opioid drug piritramide delivered via Patient-Controlled-Analgesia pump, registered daily until the 3rd postoperative day

SECONDARY OUTCOMES:
Total amount of ibuprofen; pain intensity measured on VAS-100 twice a day; Insall knee function score; incidence of analgesia side-effects ; inflammation and wound healing parameters; credibility of patients' and research stuff blinding

CONTACTS AND LOCATIONS:
Overall Officials: Hardy Edinger, Resident in Anesth, Principal Investigator — Anesthesiology and Intensive Care Medicine Department, Ernst Moritz Arndt University of Greifswald, Germany
Locations (1):
- Anesthesiology and Intensive Care Medicine Department, University of Greifswald, Germany, Greifswald, Germany

REFERENCES:
- [Result] Usichenko TI, Edinger H, Witstruck T, Pavlovic D, Zach M, Lange J, Gizhko V, Wendt M, Koch B, Lehmann C. Millimetre wave therapy for pain relief after total knee arthroplasty: a randomised controlled trial. Eur J Pain. 2008 Jul;12(5):617-23. doi: 10.1016/j.ejpain.2007.10.004. Epub 2007 Nov 26. PMID 18042413